CLINICAL TRIAL: NCT00421915
Title: Multicenter, Double-Blind, Parallel, Placebo-Controlled, Randomised Phase 3 Study of Etanercept in the Treatment of Patients With Ankylosing Spondylitis: 12-Week Final Data
Brief Title: Study Evaluating Etanercept Treatment of Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-311
Record Dates: First submitted 2007-01-08; First posted 2007-01-15 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

INTERVENTIONS:
Drug: Enbrel (etanercept)

SUMMARY:
The primary objective of the study was to compare the efficacy of etanercept (25 mg, twice weekly) with that of placebo based on the percentage of patients who achieve the Assessment in Ankylosing Spondylitis (ASAS) response criteria (ASAS 20%) at week 12.

ELIGIBILITY:
Main inclusion criteria

* Diagnosis of AS (defined by Modified New York Criteria for Ankylosing Spondylitis).
* Active AS (defined by the average of scores on the visual analog scale [VAS] of ≥ 30 for duration and intensity of morning stiffness and by 2 of the following: VAS for patient global assessment ≥ 30; average of VAS for nocturnal and total pain ≥ 30; BASFI ≥ 30 (all scores on a scale of 0 to 100).
* 18 to 70 years of age.

Main exclusion criteria

* Complete ankylosis (fusion) of spine.
* Previous receipt of etanercept, antibody to tumour necrosis factor alpha (TNFα), or other TNFα inhibitors.
* Use of disease-modifying antirheumatic drugs (DMARDs) other than hydroxychloroquine, sulphasalazine, or methotrexate within 4 weeks of baseline.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2002-03; Study Completion 2002-08

PRIMARY OUTCOMES:
To compare the efficacy of etanercept (25 mg, twice weekly) with that of placebo based on the
percentage of patients who achieved the assessment in Ankylosing Spondylitis (ASAS 20%) response criteria at week 12.

SECONDARY OUTCOMES:
To assess: 1) the safety of etanercept in this patient population; 2) the efficacy of etanercept
compared with that of placebo using the ASAS response criteria at 50% and 70% levels at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Baraliakos X, Szumski AE, Kwok KK, Vlahos B, Borlenghi CE. Long-term Etanercept Response for Patients with Radiographic Axial Spondyloarthritis Based on Achievement of Early, Intermediate, or Late Responses During Index Studies. Rheumatol Ther. 2024 Jun;11(3):583-597. doi: 10.1007/s40744-024-00656-3. Epub 2024 Mar 15. PMID 38488976
- [Derived] Baraliakos X, Szumski A, Koenig AS, Jones H. The role of C-reactive protein as a predictor of treatment response in patients with ankylosing spondylitis. Semin Arthritis Rheum. 2019 Jun;48(6):997-1004. doi: 10.1016/j.semarthrit.2018.10.019. Epub 2018 Nov 2. PMID 30473179